CLINICAL TRIAL: NCT03109860
Title: Can the Perception of a Treatment Influence Pain Processing - an Examination of Psychological and Neurobiological Mechanisms
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: The Augustinus Foundation, Denmark. (Other); The (Danish) Foundation for Neurological Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: Ina
Record Dates: First submitted 2017-04-05; First posted 2017-04-12 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-04

CONDITIONS: Neuropathic Pain
Keywords: Chronic neuropathic pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Open-hidden — Administration of a treatment openly (in full view of the patient) vs hidden (without the patient's knowledge).

SUMMARY:
The study investigates the effect of an open (in full view of the patient) vs hidden treatment (without the patient's knowledge).

ELIGIBILITY:
Inclusion Criteria:

- Neuropathic pain > 3 on a 0-10 NRS.

Exclusion Criteria:

* Psychiatric or competing neurological disorders.
* Known allergies to any medications, including local anesthetics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic neuropathic pain after thoracic surgery.
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2015-04-17 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Mechanical visual analogue scale | 10 minutes after treatment administration
  Neuropathic pain assessed on mechanical visual analogue scale

IPD SHARING:
Plan to Share IPD: No